CLINICAL TRIAL: NCT01871922
Title: Evaluation of the Effects of the Addition of Atropine During Propofol/Remifentanil Induction of Anesthesia on Hemodynamics, Microvascular Blood Flow and Tissue Oxygenenation in Patients Undergoing Ophthalmic Surgery
Brief Title: Atropine-effect During Propofol/Remifentanil Induction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Retro-002
Record Dates: First submitted 2013-05-30; First posted 2013-06-07 (Estimated); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Anesthesia-induced Negative Hemodynamic Effects
MeSH Terms: interventions — Sodium Chloride; Atropine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- General anesthesia + placebo (Placebo Comparator): Propofol/remifentanil anesthesia + saline
  Interventions: Drug: Placebo
- General anesthesia + atropine (Active Comparator): Propofol/remifentanil anesthesia + atropine
  Interventions: Drug: Atropine

INTERVENTIONS:
Drug: Placebo — Saline
  Other Names: Saline
  Arms: General anesthesia + placebo
Drug: Atropine — Atropine
  Arms: General anesthesia + atropine

SUMMARY:
Remifentanil is a widely used potent intravenous opioid with the advantage of having a short time of action. Compared to other opiates however remifentanil generates more intense hemodynamic side-effects. In ophthalmic surgery the specific anesthesiological challenges necessitate the administration of a combination of relatively high doses of analgesics on the one hand and a short time for postoperative recovery from anesthesia on the other. For these reasons, anesthetic management often consists of a combination of relatively high doses of propofol and remifentanil. A primary concern during this deep propofol/remifentanil anesthesia is preserving hemodynamic stability and adequate tissue oxygenation. Previous research of the investigators group has revealed that atropine has an exceptionally beneficial effect on hemodynamics as well as on tissue oxygenation. Therefore, the investigators hypothesize that administration of intravenous atropine during induction of propofol/remifentanil may have a positive effect on the hemodynamic profile and peripheral and cerebral tissue oxygenation during and after induction of anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring general anaesthesia;
* Patient's age ≥ 18 years and older;
* Patient and surgical procedure appropriate for treatment with either sufentanil or remifentanil.

Exclusion Criteria:

* Patient's refusal;
* Pregnancy;
* Patient's age < 18 years;
* Patients in which atropine is contra-indicated, such as severe aortic valve stenosis, hypertrophic cardiomyopathy or coronary artery disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-10; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Cardiac output | During anesthesia
Peripheral tissue oxygen saturation | During anesthesia
Cerebral tissue oxygen saturation | During anesthesia

SECONDARY OUTCOMES:
Heart rate | During anesthesia
Mean arterial blood pressure | During anesthesia
Systemic vascular resistance | During anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Alain F Kalmar, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Derived] Poterman M, Scheeren TWL, van der Velde MI, Buisman PL, Allaert S, Struys MMRF, Kalmar AF. Prophylactic atropine administration attenuates the negative haemodynamic effects of induction of anaesthesia with propofol and high-dose remifentanil: A randomised controlled trial. Eur J Anaesthesiol. 2017 Oct;34(10):695-701. doi: 10.1097/EJA.0000000000000639. PMID 28403018